

## Multi-Drug Resistant Organism Network (MDRO NETWORK)

Protocol Name: MDRO Network

Funding Sponsor: Antibiotic Resistance Leadership Group (ARLG)

Trial Identifier and Registry Name: NCT03646227

Funding Mechanism: This project is funded by the National Institute of Allergy and Infectious Diseases of the National Institutes of Health under Award Number UM1AI104681

Protocol Date: 31 August 2018

Protocol Version: Version 3.0

Study Sponsor: ARLG

Principal Investigator: David van Duin, MD, PhD

Associate Professor of Medicine Division of Infectious Diseases University of North Carolina



#### **SIGNATURE PAGE**

The signature below documents the review and approval of this protocol and provides the necessary assurances that this study will be conducted according to the protocol, including all statements regarding confidentiality, and according to national, regional, and local legal and regulatory requirements.

| Site Principal Investigator Name (Print) | <u> </u> |
|------------------------------------------|----------|
| Signature | Date |



#### **MDRO Network – Study Contact Information:**

#### Protocol Chair and Principal Investigator

David van Duin, MD, PhD Associate Professor of Medicine Division of Infectious Diseases University of North Carolina

#### Co-Principal Investigator

Robert A. Bonomo, MD Professor of Medicine, Pharmacology, Molecular Biology and Microbiology Chief, Medical Service Louis Stokes Cleveland Department of Veterans Affairs Medical Center University Hospitals Case Medical Center

#### **Coordinating Center**

The coordinating center for the MDRO Network will be Duke Clinical Research Institute. Dr. van Duin is the Principal Investigator (PI) and will be directly overseeing all activities.

#### **ARLG Publication Committee**

The ARLG Publication Committee comprises representatives of the network cores, thought-leaders, and the ARLG Statistical and Data Management Center (SDMC), and is responsible for generation and coordination of the publications that report scientific findings of the network.



# **List of Abbreviations**

| ARLG | Antibacterial Resistance Leadership Group |
|---|---|
| BSI | Bloodstream infection |
| CDC | Centers for Disease Control and Prevention |
| DCRI | Duke Clinical Research Institute |
| eCRF | Electronic case report form |
| FDA | Food and Drug Administration |
| GEE | Generalized estimating equation |
| ICH | International Council on Harmonisation |
| ICMJE | International Committee of Medical Journal Editors |
| ICU | Intensive Care Unit |
| IDES | Internet Data Entry System |
| MDRO | Multi-Drug Resistant Organism |
| IRB | Institutional Review Board |
| MALDI-TOF | Matrix-assisted laser desorption ionization time of flight mass spectrometry |
| MIC | Minimum inhibitory concentration |
| MLST | Multilocus sequence typing |
| NIAID | National Institutes of Allergy and Infectious Disease |
| NIH | National Institutes of Health |
| PBS | Pitt bacteremia score |
| PI | Principal Investigator |
| RIFLE | Risk, Injury, Failure, Loss of kidney function, and End-stage kidney disease |
| SDMC | ARLG Statistical and Data Management Center |
| SOP | Standard operating procedures |
| UTI | Urinary tract infection |



# **Protocol Summary**

| Protocol Title: | Multi-Drug Resistant Organism Network - MDRO |
|---|---|
| Study Design: | Master protocol for prospective, multicenter, observational cohort studies |
| Study Population: | Hospitalized patients with multi-drug resistant organisms |
| Number of subjects: | To be specified in each study sub-protocol as outlined in Appendices |
| Clinical Samples: | Multi-drug resistant organism isolates from specimens obtained from any anatomic site |
| Estimated Start of Enrollment: | Second quarter of 2016 |
| Estimated Time to Completion: | Second quarter of 2019 |



## 1 TABLE OF CONTENTS

| M | DRO | NETWORK – STUDY CONTACT INFORMATION: | 3 |
|---|---|---|---|
| LIS | ST OF | ABBREVIATIONS | 4 |
| PF | ROTO | COL SUMMARY | 5 |
| 1 | TAB | BLE OF CONTENTS | 6 |
| 2 | BAC | CKGROUND AND RATIONALE | 8 |
| 3 | OBJ | JECTIVE | 9 |
| | 3.3 | AIM 1. IDENTIFICATION OF TARGET POPULATION AND HIGH VOLUME CENTERS | 10<br>ND |
| 4 | STU | JDY SETTING | 10 |
| 5 | STU | JDY POPULATION | 10 |
| | 5.1<br>5.2 | Inclusion Criterion | |
| 6 | STU | JDY DESIGN | 11 |
| | 6.1<br>6.2<br>6.3<br>6.4 | Overall Strategy Clinical Variables Clinical Definitions Participant Enrollment and Follow-up | 11<br>11 |
| 7 | STA | ATISTICAL ANALYSIS | 12 |
| • | 7.1<br>7.2<br>7.3 | SAMPLE SIZE ESTIMATE PRIMARY ANALYSIS TIMING OF ANALYSES | 12<br>13 |
| 8 | | IICS AND REGULATORY CONSIDERATIONS | |
| | 8.1<br>8.2 | ETHICAL STANDARDS | |
| 9 | QUA | ALITY CONTROL AND QUALITY ASSURANCE | 14 |
| 10 | DAT | TA COLLECTION, MANAGEMENT, AND ANALYSIS | 14 |
| | 10.2 | Data Management Responsibilities Data Capture Methods Study Record Retention | 15 |
| 11 | PUE | BLICATION POLICY | 15 |
| | 11.1 | Study Findings | 15 |



| 12 | 2 REFERENCES: | . 17 |
|---|---|---|
| Α | PPENDIX I: | . 18 |
| LI | ST OF ABBREVIATIONS | . 18 |
| 1 | BACKGROUND | . 18 |
| 2 | OBJECTIVE AND PRIMARY AIMS | . 18 |
| | <ul> <li>2.1 AIM 1. IDENTIFICATION OF TARGET POPULATION AND HIGH VOLUME CENTERS</li> <li>2.2 AIM 2. PROVIDE DATA ON IMPACT OF POTENTIAL INCLUSION/EXCLUSION CRITERIA ON ENROLLMENT IN FUTURE TRIALS</li> <li>2.3 AIM 3. PROVIDE DATA ON EXPECTED OUTCOMES OF PATIENTS WITH CRE INFECTIONS FOR POWER AND SAMPLE SIZE CALCULATIONS FOR FUTURE TRIALS</li> </ul> | . 19 |
| 3 | LABORATORY ASSESSMENTS | . 19 |
| 4 | EXPLORATORY AIMS | . 19 |
| | 4.1 EXPLORATORY AIM 1. THE ASSOCIATION BETWEEN BACTERIAL CHARACTERISTICS AND CLINICAL OUTCOME. PATIENTS WITH CRE | . 19<br>. 19<br>RE |
| 5 | STUDY POPULATION | . 20 |
| 6 | CLINICAL DEFINITIONS | . 20 |
| 7 | STATISTICAL ANALYSIS PLAN | . 21 |
| | 7.1 Sample Size Estimate | . 21 |
| Α | PPENDIX II: | . 22 |
| LI | ST OF ABBREVIATIONS | . 22 |
| 1 | BACKGROUND | . 22 |
| 2 | OBJECTIVE | . 22 |
| | 2.1 AIM 1. IDENTIFICATION OF TARGET POPULATION AND HIGH VOLUME CENTERS | ง<br>. <b>2</b> 3 |
| | 2.3 AIM 3. PROVIDE DATA ON EXPECTED OUTCOMES OF PATIENTS WITH CRAB INFECTIONS FOR POWER AND SAMPLE SIZE CALCULATIONS FOR FUTURE TRIALS | |
| 3 | EXPLORATORY AIMS: | . 23 |
| 4 | ENROLLMENT TARGET | . 23 |
| 5 | STUDY POPULATION | . 23 |
| 6 | CLINICAL DEFINITIONS | . 24 |
| 7 | STATISTICAL ANALYSIS PLAN | . 24 |



| | 7.1 Sample Size Estimate | . 24 |
|---|---|---|
| A | APPENDIX III: | . 25 |
| LI | IST OF ABBREVIATIONS | . 25 |
| 1 | BACKGROUND | . 25 |
| 2 | 2 OBJECTIVE | . 25 |
| | 2.1 AIM 1. TO ASSEMBLE A MULTICENTER PROSPECTIVE COHORT OF PATIENTS WITH VRE BSIs TO PROVIDE DATA ON OUTCOMES OF PATIENTS WITH VRE BSIs FOR SAMPLE SIZE CALCULATIONS FOR FUTURE TRIALS | . 26<br>1ENT |
| 3 | | |
| | THE MOLECULAR EPIDEMIOLOGY OF INFECTING ORGANISMS FOR FUTURE STUDIES | |
| 4 | | |
| 5 | | |
| 6 | CLINICAL DEFINITIONS | . 26 |
| 7 | REFERENCES | . 27 |
| A | APPENDIX IV: | . 28 |
| LI | IST OF ABBREVIATIONS | . 28 |
| 1 | BACKGROUND | . 28 |
| 2 | OBJECTIVES | . 28 |
| | 2.1 AIM 1 2.2 AIM 2 | |
| 3 | B ENROLLMENT TARGET | . 29 |
| 4 | STUDY POPULATION | . 29 |
| | 4.1 INCLUSION CRITERIA | |
| 5 | CLINICAL DEFINITIONS | . 29 |
| 6 | STATISTICAL ANALYSIS PLAN | . 29 |
| | 6.1 Sample Size Estimate | . 29 |
| 7 | REFERENCES | . 29 |

#### 2 BACKGROUND AND RATIONALE

Per the World Health Organization, antimicrobial resistance is "one of the greatest threats to human health worldwide". In the US, infections caused by multi-drug resistant organisms (MDRO) add between \$21 billion and \$34 billion to health care costs annually, as compared to susceptible pathogens (2). In many bacterial pathogens, resistance has been increasing over the last few decades and as a general rule



clinically relevant resistance against any specific novel antibacterial either precedes or relatively quickly follows the introduction of the antibacterial for clinical use ((1), figure of timeline).



Antibiotic resistance observed

In addition to increased healthcare costs, infections with MDRO have been linked to worse patient outcomes including increased mortality (3). The study of the treatment and diagnosis of patients with MDRO infections is limited by a number of factors. First, patients with MDRO infections tend to be more chronically and acutely ill as compared to their counterparts infected with more susceptible organisms. This results in an added difficulty in prospective enrollment of these patients. Second, evaluation of outcomes in patients with MDRO infections may be complicated by a high rate of poor clinical outcomes unrelated to the infection (4). For instance, mortality unrelated to infection is unlikely to be impacted by a different antibiotic treatment strategy or an earlier diagnosis. Third, use of concomitant antibiotics prior to diagnosis of the MDRO infection is extremely common in these populations which in turn further limits enrollment into trials with restrictions on such prior treatment.

This study is specifically designed to provide data which can help in the design of future randomized clinical trials on both therapeutics and diagnostics, and describe, on the basis of observational data, patients with MDRO infections in hospitalized patients. These data will include a detailed clinical and epidemiological description of patients including potential barriers to enrollment in future trials. In addition, data will be collected on species, strain type, and mechanism of drug resistance of the causative organism. Knowing the molecular characteristics will further inform future trial design as not all diagnostics detect and not all therapeutics are active against the same mechanisms of resistance (5).

#### 3 OBJECTIVE

The objective of this study is to provide observational data that will aid in the design of randomized clinical trials on therapeutics and diagnostics for MDRO infections. To this end, clinical and epidemiological data will be collected on patients who have MDRO isolated from clinical cultures during hospitalization as well as descriptions of the outcomes of patients treated with various antimicrobial regimens. Molecular and microbiological characterization will also be performed on MDRO isolates.



#### 3.1 Aim 1. Identification of target population and high volume centers

The prevalence of specific MDRO is extremely variable in various patient populations. In addition, over time, prevalence patterns for specific MDRO tend to change. The data collection carried out under this protocol will provide real-time data on which patients are the target population for any trial directed against MDRO infection. Also, the data collected will indicate which geographic areas and which centers have the highest incidence of MDRO infections. This will facilitate rational site selection for future trials.

# 3.2 Aim 2. Provide data on impact of potential inclusion/exclusion criteria on enrollment in future trials

Detailed clinical data will be collected to guide the future development of clinical trials. The eCRF is designed to collect data on the most common barriers to enrollment in clinical trials. Data can then be used in the design of future trials to be presented to pharmaceutical companies, as well as to regulators from the FDA, to provide a rationale for requesting exceptions in inclusion/exclusion criteria. This will result in clinical trials that are more readily generalizable.

# 3.3 Aim 3. Provide data on expected outcomes of patients with MDRO infections for power and sample size calculations for future trials

In the MDRO network, detailed outcomes data will be collected. Data will include survival and microbiologic clearance outcomes when available. In addition, anatomical site specific clinical symptomatic outcomes, modeled on FDA guidance documents, will be documented. Data obtained will aid in guiding the design of future clinical trials by providing data needed for power and sample size calculations.

#### 4 STUDY SETTING

Study sites from across all five regions of the continental US and international sites from multiple countries will participate in the MDRO Network.

#### 5 STUDY POPULATION

Cohorts will be constructed for each MDRO of eligible patients by investigating hospitalized patients who have an MDRO isolated in clinical cultures from any anatomical site. This study will be conducted under a waiver of informed consent to facilitate universal inclusion. All patients who are admitted to one of the participating hospitals and who have a MDRO – as defined in the specific sub-study protocol (Appendices) – isolated in a clinical culture are targeted for inclusion.

#### 5.1 Inclusion Criterion

All hospitalized patients, including pediatric patients, who have at least one MDRO – as defined in the MDRO specific Appendices – isolated from a clinical culture will be eligible for inclusion.

#### 5.2 Exclusion Criterion

Patients who only have a positive culture for MDRO- as defined in the MDRO specific Appendices – that is obtained outside the hospital setting and do not have a positive



culture for MDRO during hospitalization.

#### **6 STUDY DESIGN**

#### 6.1 Overall Strategy

The MDRO Network will enroll at multiple sites globally. For each patient identified as having an MDRO, the data manager at the site will access the patient's medical record and use web-based data entry to enter the relevant data into the electronic case report form (eCRF) for the study's centralized database.

All MDRO isolates will be sent to the central research laboratories for molecular and microbiologic analysis. Molecular and microbiologic analyses may include, but will not be limited to, antimicrobial susceptibility testing, determination of mechanisms of antibiotic resistance, and strain typing.

#### 6.2 Clinical Variables

At both enrollment and then at 90 days after discharge from the index hospitalization during which MDRO was identified, a limited data set will be collected for each patient, and entered into a secure database. Patient demographics and co-morbid conditions; antibiotic allergies; length of hospital stay prior to first positive culture; ICU stay; reason for hospitalization; complications during hospitalization such as renal failure; components of the Pitt Bacteremia Score and Charlson comorbidity index; anatomic site-specific risk factors such as lines and devices; antibiotic use; and outcomes including all-cause and attributable mortality will be included. Specific data will be collected based on the anatomical site from which MDRO was isolated; data will include relevant symptomatology, radiographic imaging results, laboratory results, and specific interventions. Length of stay after isolation of MDRO, disposition, and readmission rates will also be collected. To specifically track the origin and spread of MDRO, detailed information regarding the origin and post-hospital disposition of each patient will be collected; for long term care facilities, the specific facility will be noted, for home origin or discharge, the first 3 digits of the international zip code will be used.

#### 6.3 Clinical Definitions

**MDRO:** Specific Multi-Drug Resistant Organisms of interest are defined in the Appendices

**Culture episode:** A positive MDRO culture from any anatomical site marks the beginning of a culture episode that includes any subsequent cultures within 7 days from the same site and during the same hospital admission. If a period of more than 7 days elapses between positive cultures, this is considered the start of a new culture episode. A positive MDRO culture from a different anatomical site is considered a separate culture episode.

**Hospital Setting:** For the purposes of this protocol, patients are considered to be in a hospital setting during the first positive MDRO culture if they are admitted to a short-term acute care hospital, or if they are in the emergency department awaiting admission with a subsequent admission. In addition, a stay in the emergency department of >24



hours will qualify as a hospital setting.

*Infection:* A patient is deemed to have an infection if a MDRO is isolated from blood or any other sterile source. For patients with positive respiratory cultures the criteria outlined by the American Thoracic Society (ATS) and the Infectious Diseases Society of America (IDSA) are used (6, 7). For patients with positive cultures from urine or surgical wounds, the CDC/National Healthcare Safety Network (NHSN) criteria are used (8). Patients with cultures from non-surgical wounds are considered infected only if the treating physician documents infection in the medical record and evidence of systemic inflammation on the day the positive culture is documented, defined as an abnormal systemic white cell count (either >10K cells/uL or <4K cells/uL), and/or abnormal body temperature (either >99.5 °F or <96 °F).

**Colonization:** All culture episodes that do not meet the preceding definitions of infection are designated as colonization (9).

**Renal failure:** Renal failure will be defined using the Risk, Injury and Failure components of the Risk, Injury, Failure, Loss of kidney function, and End-stage kidney disease RIFLE criteria (10).

**Severity of acute illness:** The Pitt bacteremia score (PBS) is calculated using temperature, mental status, cardiac arrest, blood pressure, mechanical ventilation, as described (11).

**Chronic comorbidity:** The Charlson Comorbidity Index will be calculated using documented history of myocardial infarct, congestive heart failure, peripheral vascular disease, cerebrovascular disease, dementia, chronic pulmonary disease, connective tissue disease, ulcer disease, liver disease, diabetes, hemiplegia, renal failure, any tumor, leukemia, lymphoma, AIDS, as described (12).

#### 6.4 Participant Enrollment and Follow-up

The demographic and hospitalization data will be entered in the eCRF once the patient is enrolled per eligibility criteria. The timing of the remaining data entry will be at 90 days after the conclusion of the index hospitalization. If a patient is readmitted to a study hospital and again meets criteria for inclusion in the study, a new enrollment episode will be created in the database.

#### 7 STATISTICAL ANALYSIS

#### 7.1 Sample Size Estimate

The estimated sample size for each MDRO is documented in the MDRO specific section of the Appendices.

#### 7.2 Primary Analysis

Data will be analyzed as outlined in each appendix. Furthermore, comparative analyses between different organisms will be performed.

The primary analysis will summarize the key clinical, epidemiologic, and molecular data



on patients with MDRO isolated from clinical cultures during hospitalization. Data will serve to determine potential eligibility for future trials. Strain data and mechanism of resistance will aid in determining the likelihood of response to novel antibiotic options, based on other *in vitro* and animal studies. 95% confidence intervals will be provided on key outcomes.

Data to be summarized include the following:

- Demographics
- Origin (skilled nursing facility, home, long term acute care facility, transfer from another hospital)
- Disposition (skilled nursing facility, home, long term acute care facility, transfer to another hospital, death, hospice)
- Charlson Score
- Pitt Bacteremia Score
- Source of positive culture (blood, respiratory, urine, wound, abdominal, other)
- Outcome (length of stay, ICU admission, discharge location, death)
- Antibiotic summary
- Status at 90 days
  - Defined as 90 days after the index culture. However, data will be collected through 90 days after discharge from index hospitalization.

#### 7.3 Timing of Analyses

Data will be analyzed approximately 3 times yearly in order to prepare data for reporting at annual meetings as well as for publication.

#### 8 ETHICS AND REGULATORY CONSIDERATIONS

#### 8.1 Ethical Standards

The procedures set forth in this study protocol are designed to ensure that the site investigators abide by International Council on Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) and Good Clinical Practice (GCP) guidelines in the conduct, evaluation, and documentation of this study.

Site Investigators agree, when signing the protocol, to adhere to the instructions and procedures described in it and thereby to adhere to the principles of GCP that it conforms to.

The investigator will ensure that the study will be conducted in accordance with all applicable national, regional, and local regulations.

This study will request a waiver of informed consent, consistent with country specific regulations. The study does not involve direct interaction with human subjects. The medical records of patients admitted to the hospital will be screened and data collected from those records according this protocol. The patients will not be approached to obtain information, no intervention is being tested nor are human specimens being



collected. Only pathogen MDRO isolates will be collected and analyzed.

#### 8.2 Data Confidentiality

Each participating site will prepare and maintain complete and accurate study documentation and research records for this study, in compliance with ICH E6 as well as applicable national, regulatory, and institutional requirements. The site investigator, in compliance with GCP standards, will for each participant in the study, promptly complete all eCRFs. The site investigator will comply with any other IRB or Ethics Committee requirements as stipulated by local regulations.

The sponsor's representative, Duke Clinical Research Institute (DCRI), will use a configured electronic data capture (EDC) RAVE database, to collect study data. Access will be limited to study personnel who are issued a unique user identification and password and are listed on the authorized study user list.

By signing the protocol, the site investigator acknowledges that, within legal and regulatory restrictions and institutional and ethical considerations, study documentation will be promptly and fully disclosed to the sponsor or their representative by the site investigator upon request and also shall be made available at the site investigator's site upon request for inspection, copying, review and audit at reasonable times by representatives of the sponsor or by responsible government agencies as required by law.

#### 9 QUALITY CONTROL AND QUALITY ASSURANCE

The DCRI will implement a Data Driven Trial Management Plan to ensure data quality.

By signing this protocol, the Sponsor agrees to be responsible for implementing and maintaining a quality management system with written procedures and standard operating procedures (SOPs) to ensure that the study is conducted and data are generated, documented, and reported in compliance with the protocol, accepted standards of Good Clinical Practice, and all applicable federal, state, and local laws, rules and regulations relating to the conduct of the study.

#### 10 DATA COLLECTION, MANAGEMENT, AND ANALYSIS

The site investigator is responsible to ensure the accuracy, completeness, legibility, and timeliness of the data reported. Data reported in the eCRF derived from source documents must be consistent; discrepancies should be explained in the comments field in the eCRF. The study team may provide guidance to site investigators on making corrections to the source documents and eCRF.

#### 10.1 Data Management Responsibilities

All source documents must be reviewed by the site data entry staff, who will ensure that they are accurate and complete. Data collection is the responsibility of the clinical study staff at the site under the supervision of the site investigator. During the study, the site investigator must maintain complete and accurate documentation for the study. The ARLG Statistical and Data Management Center (SDMC) will serve as the statistical and data coordinating center for this study and will be responsible for data management, quality review, analysis, and reporting of the study data.



#### 10.2 Data Capture Methods

Clinical and laboratory data will be entered into a Web-based Internet Electronic Data Capture System (EDC) that ensures data confidentiality. The data system includes individual user accounts with password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate. Clinical data will be entered directly from the source documents.

#### 10.3 Study Record Retention

Study documents should be retained per local regulations or 6 years after the end of the study, whichever is longer. No records will be destroyed without the written consent of the sponsor. It is the responsibility of the sponsor to inform the site investigator when these documents no longer need to be retained.

#### 11 PUBLICATION POLICY

#### 11.1 Study Findings

The principal investigator may publish the results of this research in a scientific journal under the oversight of the MDRO Network and ARLG Publication Committees.

The ARLG Publication Committee comprises representatives of the network cores, thought leaders, and the SDMC, and is responsible for generation and coordination of the publications that report scientific findings of the network. All public presentations (abstracts, manuscripts, slides and text of oral or other presentations, and text of any transmission through any electronic media) by participating investigators, participating institutions, the SDMC, and ARLG that use ARLG data and are intended to represent the ARLG or are supported by the ARLG will be reviewed by the Publication Committee per the Publication Committee charter and must include the following statement "Research reported in this publication was supported by the National Institute Of Allergy And Infectious Diseases of the National Institutes of Health under Award Number UM1AI104681 (The Antibacterial Resistance Leadership Group – ARLG). The content is solely the responsibility of the authors and does not necessarily represent the official views of the National Institutes of Health."

The Publication Committee guarantees that the study results are presented by experts in the field who have working knowledge of the study design, implementation, data synthesis/analysis, and interpretation. The committee goals are to ensure that any confidential or proprietary information is protected, and that all appropriate statistical analyses have been included.

All investigators funded by the NIH must submit or have submitted for them to the National Library of Medicine's PubMed Central an electronic version of their final, peer-reviewed manuscripts upon acceptance for publication, to be made publicly available no later than 12 months after the official date of publication. The NIH Public Access Policy ensures the public has access to the published results of NIH-funded research. It requires investigators to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive PubMed Central upon acceptance for publication. Further, the policy stipulates that these papers must be accessible to the public on PubMed Central no later than 12 months after publication. Refer to:



# http://publicaccess.nih.gov



#### 12 REFERENCES:

- 1. **Clatworthy AE, Pierson E, Hung DT.** 2007. Targeting virulence: a new paradigm for antimicrobial therapy. Nat Chem Biol **3:**541-548.
- 2. Spellberg B, Blaser M, Guidos RJ, Boucher HW, Bradley JS, Eisenstein BI, Gerding D, Lynfield R, Reller LB, Rex J, Schwartz D, Septimus E, Tenover FC, Gilbert DN. 2011. Combating antimicrobial resistance: policy recommendations to save lives. Clin Infect Dis 52(Suppl 5):S397-428.
- 3. **Vardakas KZ, Rafailidis PI, Konstantelias AA, Falagas ME.** 2013. Predictors of mortality in patients with infections due to multi-drug resistant Gram negative bacteria: the study, the patient, the bug or the drug? J Infect **66:**401-414.
- 4. Hauck C, Cober E, Richter SS, Perez F, Salata RA, Kalayjian RC, Watkins RR, Scalera NM, Doi Y, Kaye KS, Evans S, Fowler VG, Jr., Bonomo RA, van Duin D, Antibacterial Resistance Leadership G. 2016. Spectrum of excess mortality due to carbapenem-resistant Klebsiella pneumoniae infections. Clin Microbiol Infect 22:513-519.
- 5. **Zasowski EJ, Rybak JM, Rybak MJ.** 2015. The beta-Lactams Strike Back: Ceftazidime-Avibactam. Pharmacotherapy **35:**755-770.
- 6. Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM, Jr., Musher DM, Niederman MS, Torres A, Whitney CG. 2007. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis 44 Suppl 2:S27-72.
- 7. **American Thoracic Society and Infectious Diseases Society of America.** 2005. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med **171:**388-416.
- 8. **Centers for Disease Control and Prevention.** January 2014 2014. CDC/NHSN Surveillance Definitions for Specific Types of Infections. www.cdc.gov/nhsn. Accessed
- 9. van Duin D, Perez F, Rudin SD, Cober E, Hanrahan J, Ziegler J, Webber R, Fox J, Mason P, Richter SS, Cline M, Hall GS, Kaye KS, Jacobs MR, Kalayjian RC, Salata RA, Segre JA, Conlan S, Evans S, Fowler VG, Jr., Bonomo RA. 2014. Surveillance of Carbapenem-Resistant Klebsiella pneumoniae: Tracking Molecular Epidemiology and Outcomes through a Regional Network. Antimicrob Agents Chemother 58:4035-4041.
- 10. **Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P, Acute Dialysis Quality Initiative w.** 2004. Acute renal failure definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care **8:**R204-212.
- 11. **Chow JW, Yu VL.** 1999. Combination antibiotic therapy versus monotherapy for gram-negative bacteraemia: a commentary. Int J Antimicrob Agents **11:**7-12.
- 12. **Charlson ME, Pompei P, Ales KL, MacKenzie CR.** 1987. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis **40:**373-383.



#### Appendix I:

CRACKLE II: Consortium on Resistance Against Carbapenems in Klebsiella pneumoniae and Other Enterobacteriaceae (CRACKLE): a Prospective, Observational Cohort Study

#### **List of Abbreviations**

| CRACKLE | Consortium on Resistance Against Carbapenems in <i>Klebsiella</i> pneumoniae and other Enterobacteriaceae |
|---|---|
| CRE | Carbapenem-resistant Enterobacteriaceae |
| CRKP | Carbapenem-resistant Klebsiella pneumoniae |
| K. pneumoniae | Klebsiella pneumoniae |
| PCR | Polymerase Chain Reaction |
| rep-PCR | Repetitive extragenic palindromic polymerase chain reaction |
| ST258 | Sequence type 258 |

#### 1 Background

Carbapenem resistance is increasingly common in Enterobacteriaceae (CRE), especially *Klebsiella pneumoniae* (*K. pneumoniae*) isolates, and represents a major threat to our global population. Since the first reported carbapenem-resistant *K. pneumoniae* (CRKP) was identified in 1996, the incidence of infections due to this multidrug-resistant (MDR) pathogen has increased dramatically. According to data from the Centers of Disease Control (CDC), 11% of K. pneumoniae that cause healthcare-associated infections are carbapenem resistant. Regrettably, outcomes after CRKP bloodstream infections are generally poor. All-cause mortality rates of 42-72% have been reported. The globally endemic CRKP strain type 258 (ST258) is responsible for the majority of infections in the US. The mechanism of resistance for most ST258 isolates in the US is the Klebsiella pneumoniae carbapenemase (KPC) family.

#### 2 Objective and Primary Aims

The objective of this study is to provide observational data that will aid in the design of randomized clinical trials on therapeutics and diagnostics for CRE infections. To this end, clinical and epidemiological data will be collected on patients who have CRE isolated from clinical cultures during hospitalization as well as descriptions of the outcomes of patients treated with various antimicrobial regimens. Molecular and microbiological characterization will also be performed on CRE isolates.



#### 2.1 Aim 1. Identification of target population and high volume centers

The prevalence of specific CRE is extremely variable in various patient populations. In addition, over time, prevalence patterns for specific CRE tend to change. The data collection carried out under this protocol will provide real-time data on which patients who are the target population for any trial directed against CRE infection. Also, the data collected will indicate which geographic areas and which centers have the highest incidence of CRE infections. This will facilitate rational site selection for future trials.

# 2.2 Aim 2. Provide data on impact of potential inclusion/exclusion criteria on enrollment in future trials

Detailed clinical data will be collected to guide the future development of clinical trials. The eCRF is designed to collect data on the most common barriers to enrollment in clinical trials. Data can then be used in the design of future trials to be presented to pharmaceutical companies, as well as to regulators from the FDA, to provide a rationale for requesting exceptions in inclusion/exclusion criteria. This will result in clinical trials that are more readily generalizable (see 3.2 in main MDRO protocol).

# 2.3 Aim 3. Provide data on expected outcomes of patients with CRE infections for power and sample size calculations for future trials

Detailed outcomes data will be collected. Data will include survival and microbiologic clearance outcomes when available. In addition, anatomical site specific clinical symptomatic outcomes, modeled on FDA guidance documents, will be documented. Data obtained will aid in guiding the design of future clinical trials by providing data needed for power and sample size calculations (see 3.3 in main MDRO protocol).

#### 3 Laboratory Assessments

As novel antibiotics directed against CRE may have differential efficacy based on the mechanism of resistance, molecular characterization for strain type and mechanism of carbapenem resistance will be performed on CRE isolates, including whole genome sequencing, single gene PCR, multilocus sequence typing (MLST) and/or rep-PCR (6). Furthermore, phenotypic characteristics such as *in vitro* susceptibility testing will be performed in the central research laboratories.

#### 4 Exploratory Aims

- 4.1 Exploratory Aim 1. The association between bacterial characteristics and clinical outcomes in patients with CRE
- 4.2 Exploratory Aim 2. The association between treatment modalities and clinical outcomes in patients with CRE
- 4.3 Exploratory Aim 3. Risk factors for baseline and treatment-emergent resistance to anti-CRE antibacterials in patients with CRE



#### 5 Study Population

All patients who are admitted to one of the participating hospitals and who have a CRE isolated from bloodstream infection source in a clinical culture will be included.

In addition, all participating hospitals in China will also enroll patients who meet the below criteria:

- a. have a CRE isolated from respiratory source in a clinical culture
- b. AND have a clinical diagnosis of pneumonia, per diagnosis criteria in Table 1

Table 1.

| | At least one criterion from each section must be present to meet definition of pneumonia diagnosis | |
|---|---|---|
| 1 | Radiographic<br>Criteria | Chest radiograph showing the presence of new or progressive infiltrate(s) suggestive of bacterial pneumonia within 48 hours of all other diagnostic criteria being present |
| 2 | Respiratory<br>Signs/Symptoms | • New onset or worsening: cough, dyspnea, tachypnea (respiratory rate >= 25 breaths per minute for patients >18 years, >60 breaths per minute for children <1 year, >40 breaths per minute for children ages 1-3 years, >30 breaths per minute for children ages 4-12 years, >20 breaths per minute for children 12-18 years), or expectorated sputum production |
| | | <ul> <li>Hypoxemia, defined as any of the following: <ul> <li>A partial pressure of oxygen &lt;60 millimeters of mercury measured by arterial blood gas (ABG)</li> <li>A worsening (decrease &gt;10%) of the ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2)</li> <li>Pulse oximetry reading of &lt;90%</li> <li>New supplemental oxygen requirement</li> <li>Greater than 2LPM increase in amount of supplemental oxygen required for patients on chronic supplemental oxygen therapy</li> <li>Need for acute changes, after 2 days stability, in ventilator support system to enhance oxygenation, as determined by worsening oxygenation (ABG or PaO2/FiO2) or needed changes in the amount of positive end-expiratory pressure</li> </ul> </li> </ul> |
| 3 | Systemic<br>Inflammation | <ul> <li>Documented body temperature ≥38 degrees Celsius or ≤ 35 degrees Celsius (core body temperature)</li> <li>Leukocytosis, defined as total peripheral white blood cell count ≥10,000 cells/cubic millimeter</li> <li>Leukopenia, defined as total peripheral white blood cell count ≤4,500 cells/cubic millimeter</li> </ul> |
| | | Greater than 15% immature neutrophils (bands) noted on peripheral blood film |

#### 6 Clinical Definitions

**CRE**: For the purposes of this study, CRE are defined as any Enterobacteriaceae displaying in vitro resistance to any of the carbapenems as per CDC guidelines, i.e. Enterobacteriaceae that are resistant to any carbapenem antimicrobial (i.e., minimum inhibitory concentrations of ≥4 mcg/ml for doripenem, meropenem, or imipenem OR ≥2



mcg/ml for ertapenem) OR Documented to produce carbapenemase.

#### In addition:

• For bacteria that have intrinsic imipenem nonsusceptibility (i.e., Morganella morganii, Proteus spp., Providencia spp.), resistance to carbapenems other than imipenem is required.

## 7 Statistical Analysis Plan

## 7.1 Sample Size Estimate

The sample size is estimated to be between 3,000-5,000 unique admissions.



#### Appendix II:

SNAP: Study Network of Acinetobacter baumannii as Carbapenem-Resistant Pathogen

#### **List of Abbreviations**

| SNAP | Study Network of <i>Acinetobacter baumannii</i> as Carbapenem-Resistant Pathogen |
|---|---|
| CRAb | Carbapenem-resistant Acinetobacter baumannii |
| PCR | Polymerase Chain Reaction |
| rep-PCR | Repetitive extragenic palindromic polymerase chain reaction |

#### 1 Background

Acinetobacter baumannii has emerged as one of the most highly antimicrobial-resistant pathogens causing hospital-acquired infections globally. In the U.S., an estimated 45,000 cases of *A. baumannii* infections occur per year. The most common presentations of invasive infection include bacteremia and pneumonia. A. baumannii has an extraordinary ability to develop resistance to even the most potent antimicrobial agents. In particular, carbapenem resistance among A. baumannii has dramatically increased in the last decade, with rates increasing from 21% in 2003-2005 to 48% in 2009-2012. According to recent CDC data, 55% of A. baumannii causing ventilatorassociated pneumonia in the U.S. are resistant to carbapenems. Treatment options for carbapenem-resistant A. baumannii (CRAb) infections are extremely limited and include agents such as colistin, tigecycline and minocycline, which have uncertain efficacy and considerable toxicity. Risk factors for acquiring CRAb include exposure to antimicrobial agents, presence of indwelling catheters, severity of illness, and length of hospital stay especially in intensive care units. In-hospital and 30-day all-cause mortality from CRAb infections are estimated to be 42%-62% and 16%-58%, respectively. Despite this significant disease burden, prospective multicenter studies that evaluate microbiological factors that impact patient outcome – while carefully controlling for clinical co-variables have not yet been conducted in the U.S.

#### 2 Objective

The objective of this study is to provide observational data that will aid in the design of randomized clinical trials on therapeutics and diagnostics for CRAb infections. To this end, clinical and epidemiological data will be collected on patients who have CRAb isolated from clinical cultures during hospitalization as well as descriptions of the outcomes of patients treated with various antimicrobial regimens. Molecular and



microbiological characterization will also be performed on CRAb isolates.

#### 2.1 Aim 1. Identification of target population and high volume centers

The prevalence of specific CRAb is extremely variable in various patient populations. In addition, over time, prevalence patterns for specific CRAb tend to change. The data collection carried out under this protocol will provide real-time data on which patients are the target population for any trial directed against CRAb infection. Also, the data collected will indicate which geographic areas and which centers have the highest incidence of CRAb infections. This will facilitate rational site selection for future trials.

# 2.2 Aim 2. Provide data on impact of potential inclusion/exclusion criteria on enrollment in future trials

Detailed clinical data will be collected to guide the future development of clinical trials. The eCRF is designed to collect data on the most common barriers to enrollment in clinical trials. Data can then be used in the design of future trials to be presented to pharmaceutical companies, as well as to regulators from the FDA, to provide a rationale for requesting exceptions in inclusion/exclusion criteria. This will result in clinical trials that are more readily generalizable (see 3.2 in main MDRO protocol).

# 2.3 Aim 3. Provide data on expected outcomes of patients with CRAb infections for power and sample size calculations for future trials

Detailed outcomes data will be collected. Data will include survival and microbiologic clearance outcomes when available. In addition, anatomical site specific clinical symptomatic outcomes, modeled on FDA guidance documents, will be documented. Data obtained will aid in guiding the design of future clinical trials by providing data needed for power and sample size calculations (see 3.3 in main MDRO protocol).

#### 3 Exploratory Aims:

- -To establish a prospective cohort of subjects with carbapenem-resistant *Acinetobacter* baumannii infection or colonization
- -To describe the demographics, natural history and clinical outcome of patients with CRAb
- -To collect the associated A. baumannii strains of patients with CRAb for future studies

#### 4 Enrollment Target

The study will enroll up to 2000 unique admissions. This will be a global competitive enrollment.

#### 5 Study Population

All patients who are admitted to one of the participating hospitals and who have a CRAb isolated in a clinical culture will be included.



#### 6 Clinical Definitions

**CRAb**: Acinetobacter baumannii isolates that are resistant (minimum inhibitory concentrations of ≥8 mcg/ml) to at least one of the following three carbapenems: doripenem, imipenem, meropenem.

## 7 Statistical Analysis Plan

## 7.1 Sample Size Estimate

The sample size will be approximately 2000 unique admissions.



#### Appendix III:

VENOUS II: Vancomycin-Resistant Enterococci Outcomes Study II

#### **List of Abbreviations**

| VENOUS II | Vancomycin-Resistant Enterococci Outcomes Study II |
|-----------|----------------------------------------------------|
| VRE | Vancomycin-Resistant Enterococci |
| BSI | Blood Stream Infection |

#### 1 Background

Vancomycin-resistant enterococci (VRE) are one of the leading causes of health-care associated infections, causing approximately 20,000 infections and 1,300 deaths per year in the US alone (1). Moreover, VRE are a major cause of bloodstream infections (BSI) and preferentially affect patients who are severely ill and have an impaired immune system, such as cancer patients and subjects in the intensive care setting (2). Currently, there is only one FDA-approved drug to treat VRE (linezolid). However, linezolid has major limitations for the treatment of severe VRE infections and its use in patients that need prolonged therapy is discouraged due to an unfavorable toxicity profile. Although several new drugs have been approved for the management of other important drug-resistant gram-positives (e.g. methicillin-resistant Staphylococcus aureus), the majority of these new compounds lack bactericidal activity against VRE. The most common anti-VRE used drug is daptomycin (off-label), a lipopeptide antibiotic with in vitro bactericidal activity against these organisms (3). However, the emergence of resistance during daptomycin therapy is a serious concern and uncertainty in the best dose regimen to treat severe VRE infections remains (4). Thus, robust clinical data to determine the best treatment approaches for these multi-drug resistant organisms are urgently needed. Indeed, despite the significant burden of disease caused by VRE, prospective multicenter studies evaluating clinical and microbiological factors that impact patient outcomes have not yet been conducted in the U.S.

## 2 Objective

The objective of this study is to establish a large multicenter prospective cohort of patients with VRE BSIs to provide solid observational data that will aid in the design of randomized clinical trials on therapeutics and diagnostics for deep-seated VRE infections. To this end, clinical and epidemiological data will be collected on patients who have VRE isolated from the bloodstream during hospitalization, as well as descriptions of the outcomes of patients treated with various antimicrobial regimens. VRE isolates will also be collected to perform molecular and genomic characterization.



# 2.1 Aim 1. To assemble a multicenter prospective cohort of patients with VRE BSIs to provide data on outcomes of patients with VRE BSIs for sample size calculations for future trials

We will leverage from an ongoing effort (VENOUS I) that has prospectively collected data from ca. 200 patients with enterococcal infections from three active centers to assemble a large multicenter cohort of patients with VRE BSIs. The data collected under this protocol will provide valuable information regarding outcomes and prognostic factors (both from the patient and isolate perspective), along with real-life data on which patients are the target population for any trial directed against invasive VRE infections. Also, we expect this cohort to help pinpoint specific geographic areas and/or centers with high incidence of VRE infections, facilitating the rational selection of sites for future trials. Data on outcomes (i.e. survival and microbiologic clearance) will aid in guiding the design of future clinical trials by providing reliable information needed for power and sample size calculations (see 3.3 in main MDRO protocol).

# 2.2 Aim 2. To provide data on the impact of potential inclusion/exclusion criteria on enrollment in future VRE trials

Detailed clinical data will be collected to guide the future development of clinical trials. The eCRF is designed to collect data on the most common barriers to enrollment in clinical trials. Data can then be used in the design of future trials to be presented to pharmaceutical companies, as well as to regulators from the FDA. The information will also be used to provide a rationale for requesting exceptions in inclusion/exclusion criteria. This valuable data will result in the design of clinical trials that are more readily generalizable (see 3.2 in main MDRO protocol).

# 3 Exploratory Aim. To collect VRE isolates causing BSIs in order to understand the molecular epidemiology of infecting organisms for future studies

All infecting VRE isolates will be collected for further microbiological, molecular and genomic characterization, as part of future studies. Bacterial genomic information will be analyzed in order to find possible genetic factors that correlate with clinical outcomes in deep-seated VRE infections.

#### 4 Enrollment Target

200 unique admissions. This will be a competitive enrollment.

#### 5 Study Population

All patients admitted to one of the participating hospitals who develop a confirmed blood stream infection due to VRE will be included in the study. In order to enroll a patient, the VRE isolate should be available for further characterization.

#### 6 Clinical Definitions

**VRE BSI**: At least one blood culture positive for vancomycin-resistant enterococci (resistance to vancomcyin will be defined by current CLSI guidelines), regardless of the Enterococcal species and of the susceptibility method used by the microbiology



laboratory.

#### 7 References

- 1. Agudelo Higuita, N.I. and M.M. Huycke, *Enterococcal Disease, Epidemiology, and Implications for Treatment*, in *Enterococci: From Commensals to Leading Causes of Drug Resistant Infection*, M.S. Gilmore, et al., Editors. 2014: Boston.
- 2. Vydra J, Shanley RM, George I, Ustun C, Smith AR, Weisdorf DJ, Young JA. Enterococcal bacteremia is associated with increased risk of mortality in recipients of allogeneic hematopoietic stem cell transplantation. Clin Infect Dis. 2012;55(6):764-70.
- 3. Britt NS, Potter EM, Patel N, Steed ME. Comparison of the Effectiveness and Safety of Linezolid and Daptomycin in Vancomycin-Resistant Enterococcal Bloodstream Infection: A National Cohort Study of Veterans Affairs Patients. Clin Infect Dis. 2015;61(6):871-8.
- 4. Britt, N.S., et al., Comparative Effectiveness and Safety of Standard-, Medium-, and High-Dose Daptomycin Strategies for the Treatment of Vancomycin-Resistant Enterococcal Bacteremia Among Veterans Affairs Patients. Clin Infect Dis, 2017. **64**(5): p. 605-613.



#### **Appendix IV:**

POP: Prospective Observational *Pseudomonas* study

#### List of Abbreviations

| POP | Prospective Observational <i>Pseudomonas</i> study |
|------|----------------------------------------------------|
| CRPA | carbapenem-resistant <i>P. aeruginosa</i> |
| BSI | Blood Stream Infection |

#### 1 Background

Pseudomonas aeruginosa infections are common in immunocompromised patients, are a leading cause of hospital-acquired infection, and are associated with poor outcomes. Treatment of *P. aeruginosa* infections is complicated by antimicrobial resistance, including resistance to carbapenems. Carbapenem resistance is especially challenging because it is often associated with resistance to multiple classes of antibiotics, leaving few therapeutic options. Novel technologies and drugs are needed to better diagnose and treat *P. aeruginosa* infections, but designing the clinical trials necessary to address this demand is challenging given the lack of detailed data on *P. aeruginosa* resistance mechanisms, clinical and molecular epidemiology, treatment, and outcomes. This proposal aims to fill this gap by providing detailed clinical and microbiologic data in carbapenem-resistant *P. aeruginosa* (CRPA) pulmonary and bloodstream infections. We believe that this study is ideal for the ARLG, as it will utilize the existing the MDRO Network, which already has similar ongoing studies in patients with carbapenem-resistant Enterobacteriaceae and carbapenem-resistant *Acinetobacter* infections.

## 2 Objectives

#### 2.1 Aim 1

Define antibiotic resistance determinants and molecular epidemiology of CRPA pulmonary and bloodstream infections within the ARLG MDRO network.

#### 2.2 Aim 2

Facilitate future interventional and diagnostic studies involving CRPA by detailing current epidemiology, treatment, and outcomes of CRPA pulmonary and bloodstream infections at potential clinical trial sites within the ARLG MDRO Network.



#### 3 Enrollment Target

The study will enroll up to 2000 unique admissions. This will be a global competitive enrollment.

#### 4 Study population

#### 4.1 Inclusion criteria

All patients at participating sites, including pediatric patients, with CRPA isolated from any clinical culture during hospitalization or within 3 days prior to hospitalization will be included in the study.

#### 4.2 Exclusion criteria

- 1. Outpatient status at the time of collection of cultures that yield CRPA and patient not admitted to the hospital for CRPA infection within 3 days of collection of the culture
- 2. Cystic fibrosis

#### 5 Clinical Definitions

**CRPA:** *Pseudomonas aeruginosa* isolates that are resistant in vitro to at least one of the following carbapenems: doripenem, imipenem, meropenem.

## 6 Statistical Analysis Plan

#### 6.1 Sample Size Estimate

The sample size will be approximately 2000 unique admissions.

#### 7 References

- Que YA, Lazar H, Wolff M, Francois B, Laterre PF, Mercier E, Garbino J, Pagani JL, Revelly JP, Mus E et al: Assessment of panobacumab as adjunctive immunotherapy for the treatment of nosocomial Pseudomonas aeruginosa pneumonia. Eur J Clin Microbiol Infect Dis 2014, 33(10):1861-1867.
- 2. Lu Q, Rouby JJ, Laterre PF, Eggimann P, Dugard A, Giamarellos-Bourboulis EJ, Mercier E, Garbino J, Luyt CE, Chastre J et al: Pharmacokinetics and safety of panobacumab: specific adjunctive immunotherapy in critical patients with nosocomial Pseudomonas aeruginosa O11 pneumonia. *J Antimicrob Chemother* 2011, 66(5):1110-1116.
- 3. Forestier C, Guelon D, Cluytens V, Gillart T, Sirot J, De Champs C: **Oral probiotic and prevention of Pseudomonas aeruginosa infections: a randomized, double-blind, placebo-controlled pilot study in intensive care unit patients**. *Crit Care* 2008, **12**(3):R69.
- 4. Nichols L, Gudmundsson S, Maki DG: Experience with cefsulodin therapy for lower respiratory tract infections caused by Pseudomonas aeruginosa in adults without cystic fibrosis or granulocytopenia. *Rev Infect Dis* 1984, 6 Suppl 3:S711-720.
- 5. Deal EN, Micek ST, Reichley RM, Ritchie DJ: Effects of an alternative cefepime dosing strategy in pulmonary and bloodstream infections caused by Enterobacter spp, Citrobacter



- freundii, and Pseudomonas aeruginosa: a single-center, open-label, prospective, observational study. *Clin Ther* 2009, **31**(2):299-310.
- 6. Luyt CE, Aubry A, Lu Q, Micaelo M, Brechot N, Brossier F, Brisson H, Rouby JJ, Trouillet JL, Combes A *et al*: Imipenem, meropenem, or doripenem to treat patients with Pseudomonas aeruginosa ventilator-associated pneumonia. *Antimicrobial agents and chemotherapy* 2014, 58(3):1372-1380.
- 7. Lu Q, Yang J, Liu Z, Gutierrez C, Aymard G, Rouby JJ, Nebulized Antibiotics Study G: **Nebulized** ceftazidime and amikacin in ventilator-associated pneumonia caused by Pseudomonas aeruginosa. *Am J Respir Crit Care Med* 2011, **184**(1):106-115.
- 8. Chow JW, Yu VL: Combination antibiotic therapy versus monotherapy for gram-negative bacteraemia: a commentary. *Int J Antimicrob Agents* 1999, **11**(1):7-12.
- 9. Charlson ME, Pompei P, Ales KL, MacKenzie CR: A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. *J Chronic Dis* 1987, 40(5):373-383.
- 10. van Duin D, Perez F, Rudin SD, Cober E, Hanrahan J, Ziegler J, Webber R, Fox J, Mason P, Richter SS *et al*: **Surveillance of carbapenem-resistant Klebsiella pneumoniae: tracking molecular epidemiology and outcomes through a regional network**. *Antimicrobial agents and chemotherapy* 2014, **58**(7):4035-4041.